CLINICAL TRIAL: NCT02633085
Title: A Retrospective, Consecutive Series, Single Surgeon Study Comparing Patient Satisfaction and Clinical Outcomes in Patients With Fixed Bearing Versus Mobile Bearing Unicompartmental Knee Arthroplasty
Brief Title: Fixed Bearing Versus Mobile Bearing Patient Satisfaction and Clinical Outcome Study
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: #002 FB vs MB
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis
Keywords: Unicompartment Knee Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fixed Bearing or Mobile Bearing UKA
  Interventions: Device: Fixed Bearing or Mobile Bearing UKA

INTERVENTIONS:
Device: Fixed Bearing or Mobile Bearing UKA — Fixed Bearing or Mobile Bearing UKA Patients who have undergone a primary Fixed Bearing or a Mobile Bearing UKA in either knee and are at a minimum 2 years post-op.
  Other Names: Zimmer Unicompartmental High Flex Knee System or Oxford Mobile Bearing

SUMMARY:
The purpose of this study is to determine if there is a patient satisfaction preference of Fixed Bearing versus Mobile Bearing Unicompartmental Knee Arthroplasty (UKA) in patients who are at a minimum two years post operative. Patient reported outcomes and expectations will be analyzed along with all retrospective chart data in patient with a Fixed Bearing or a Mobile Bearing UKA in one or both knees.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to read, understand and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF)
2. Ability to understand and provide written authorization for use and disclosure of personal health information.
3. Subject who are able and willing to comply with the study protocol and follow-up visit.
4. Must be 18 years or older to participate.
5. Subjects must have a clinically documented Osteoarthritis in a knee, single or multiple compartments,
6. Subjects must have undergone a FB UKA or MB UKA in one and or both knees. MB UKA or FB UKA patients revised to Total Knee Arthroplasty (TKA) are eligible to enroll.
7. Must be a minimum 2 year (24 months) post-surgery on the knee.
8. The UKA operation must have been performed by the Investigator.
9. Subjects must be able to return for the follow-up appointment, and have the mental capacity to cooperate with PRO's, questionnaires, physical exam and imaging studies.

Exclusion Criteria:

1. Subjects with Bicompartmental UKA (i.e. medical or lateral UKA combined with Patello Femoral Joint (PFJ) (UKA)
2. Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone a Unicompartment Knee Replacement with a Fixed Bearing or Mobile Bearing prosthesis.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
To compare patient satisfaction scores of the Unicompartmental Fixed Bearing (FB) UKA vs Unicompartmental Mobile Bearing (MB) UKA | Minimum of two years post-surgery.
  Utilizing Knee Score Society survey sub-score

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Minimum of two years post-surgery.
  Knee symptoms, pain, function and Qol
Forgotten Joint Score (FJS) | Minimum of two years post-surgery.
  Knee Function-patients ability to forget the artificial joint in everyday life
Knee Society Score (KSS) subjective measures | Minimum of two years post-surgery.
  patient expectation and satisfaction sub-scores
Euro-Qual Health related Quality of Life | Minimum of two years post-surgery.
  General Health Status
Return to Work History | Minimum of two years post-surgery.
  Questionnaire for work history prior to surgery and after surgery
Radiographic Analysis | Minimum of two years post-surgery.
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Knee Society Score (KSS) Objective Measures | Minimum of two years post-surgery.
Demographics | Minimum of two years post-surgery.
Complications | Minimum of two years post-surgery.
  Complications will be recorded

OTHER OUTCOMES:
Sub-Study 1: Fixed Bearing Meta-analysis | Minimum of two years post-surgery.
  Full Knee Society Score (KSS) and Short Form Health Survey SF-12
Sub Study 2: Prosthesis positing versus outcomes analysis | Minimum of two years post-surgery.
  CT scan of Fixed Bearing patients for implant position

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Ahuja, MBBS, MS, Study Director — Medacta USA, Inc.
Locations (1):
- Tri County Orthopeadic Center, Leesburg, Florida, United States